CLINICAL TRIAL: NCT01737463
Title: Prophylactic Pancreatic Duct Stent Placement After Endoscopic Snare Papillectomy of Duodenal Major Papillary Tumors; Prospective, Randomized, Controlled Study
Brief Title: Prophylactic Pancreatic Duct Stent Placement After ESP of Major Papillary Tumors; Prospective, Randomized Study
Acronym: PDS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, Byung Hoo Lee, SoonchunhyangUH, Soonchunhyang University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MD-2012-04
Record Dates: First submitted 2012-11-16; First posted 2012-11-29 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-12

CONDITIONS: Ampulla of Vater Adenoma
Keywords: Ampulla of Vater adenoma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Active Comparator): Endoscopic snare papillectomy (ESP) was performed by using diagnostic or therapeutic duodenoscope (JF-240, TJF-240, JF-260, TJF-260; Olympus Optical Co, Ltd, Tokyo, Japan).
  A pancreatic duct stent was inserted immediately after the excision.
  Interventions: Procedure: Endoscopic snare papillectomy
- Group B (Active Comparator): Endoscopic snare papillectomy (ESP) was performed by using diagnostic or therapeutic duodenoscope (JF-240, TJF-240, JF-260, TJF-260; Olympus Optical Co, Ltd, Tokyo, Japan).
  A pancreatic duct stent was not inserted immediately after the excision.
  Interventions: Procedure: Endoscopic snare papillectomy

INTERVENTIONS:
Procedure: Endoscopic snare papillectomy — Endoscopic snare papillectomy (ESP) was performed by using diagnostic or therapeutic duodenoscope. A pancreatic duct stent was or was not inserted immediately after the excision.

SUMMARY:
Endoscopic snare papillectomy (ESP) is an efficient treatment for benign tumors of the duodenal major papilla. But post-ESP pancreatitis is the most common and serious complication. Since one prospective randomized controlled trial showed that pancreatic duct stent placement reduced post-ESP pancreatitis, almost physicians have tried to place the pancreatic duct stent after EPS.

The aim of this prospective, randomized, multicenter trial is to compare the rates of post-ESP pancreatitis in patients who did or did not prophylactic pancreatic duct stent placement. Consecutive patients who were to undergo ESP were to randomized to pancreatic duct stent placement group (stent group) after endoscopic snare papillectomy or to no pancreatic duct stent placement group (no stent group).

DETAILED DESCRIPTION:
The patient was adequately sedated by intravenous administration of midazolam with or without meperidine. ESP and pancreatic duct stent insertion were undertaken using two methods: conventional and wire-guieded ESP. The conventional ESP method was performed as in the follows. After placing the tip of the duodenoscope on the tumor, the snare was deployed so that it grasped the base of the tumor. Constant tension was applied to the snare loop during excision until the lesion was transected. Excision was performed with a small sized electrosurgical snare. A pancreatic duct stent was or was not inserted immediately after the excision. The wire-guided ESP method was performed as follows. An ERCP catheter was inserted into the pancreatic duct. Then, a 0.035-inch guidewire was inserted through the catheter and deep into the main pancreatic duct. After the ERCP catheter was removed, the loop of an electrosurgical snare with a maximum sheath diameter of 1.8 mm was passed over the guidewire, in monorail fashion, and the snare was closed lightly. The snare was introduced next to the guidewire into the accessory channel of the duodenoscope. After the tip of the duodenoscope was placed on the tumor, the snare was deployed so that it grasped the base of the tumor. Constant tension was applied to the snare loop during excision until the lesion was transected. After the excision was completed, a pancreatic duct stent was immediately passed over the guidewire previously placed in the pancreatic duct and was positioned across the pancreatic-duct oriﬁce. ESP was performed by using the blend mode or endocut mode setting on the electrosurgical generator. A straight or single pigtail type, 3- to 9-cm, 3 to 7F polyethylene pancreatic duct stent was used. Post-papillectomy bleeding was treated with argon plasma coagulation (APC) and/or endoscopic clipping or epinephrine injection. APC was carried out with a power setting of 60 W and a gas flow of 2 L/min. One to seven days after stent placement, a plain abdominal radiograph was obtained to determine its position. If it had not passed spontaneously, it was removed endoscopically from those patients with no evidence of pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20 to 80 years, Histopathologically proven ampullary adenoma

Exclusion Criteria:

* Lesions with irregular margin, ulceration and spontaneous or easy to bleeding which presenting malignancy.
* Extensive lesion into PD or BD on ERCP, EUS or IDUS.
* Tumor size > 4cm
* Bleeding tendency

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-03; Primary Completion 2013-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Prophylactic pancreatic duct stent placement after endoscopic snare papillectomy of duodenal major papillary tumors; prospective, randomized, controlled study | after October 1, 2012 (up to 2 years)
  The incidence of post-ESP pancreatitis and hyperamylasemia

SECONDARY OUTCOMES:
Prophylactic pancreatic duct stent placement after endoscopic snare papillectomy of duodenal major papillary tumors; prospective, randomized, controlled study | after October 1, 2012 (up to 2 years)
  The incidence of post-ESP pancreatitis, hyperamylasemia and post-ESP pancreatitis risk factors was compared between the groups.

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Woo Cha, PhD, Study Chair — Institute for Digestive Research, Digestive Disease Center, Department of Internal Medicine, Soonchunhyang University College of Medicine, Seoul, Korea.
Locations (1):
- Institute for Digestive Research, Digestive Disease center, Department of Internal Medicine, Soonchunhyang University College of Medicine, Yongsan-gu, Seoul, South Korea